CLINICAL TRIAL: NCT07236060
Title: Placenta Accreta Spectrum VS Uterine Scar Dehiscence: Accurate Ultrasound Model in 3rd Trimester Pregnancies for Percise Diagnosis
Brief Title: Ultrasound Model to Help Differentiate Between Placenta Accreta Spectrum and Uterine Dehiscence in 3rd Trimester Pregnancies
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Ahmed Mohammed Refaat Askalany, Resident, Assiut University
Other Study IDs: 042025201333
Record Dates: First submitted 2025-09-30; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Placenta Accreta, Third Trimester; Uterine Scar Dehiscence
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: 2D ultrasound doppler — using 2d ultrasound doppler to form a model that will help distinguish between placenta accreta spectrum and uterine scar dehiscence pre-operatively

SUMMARY:
By using 2d Ultrasound on 3rd trimester pregnant women, a model is made to help differentiate between placenta accreta spectrum and uterine scar dehiscence before operative action to help prepare multi-disciplinary steps if needed

DETAILED DESCRIPTION:
A cross-sectional observational study

ELIGIBILITY:
Inclusion Criteria:

* Women in 3rd trimester pregnancy with low lying placenta previa
* History of 1 or more C-section
* Patients planning to deliver baby in Assiut women health hospital
* Willing and able to participate

Exclusion Criteria:

* Antepartum Hemorrhage(sever attack) as it hinders time for accurate diagnosis and calling expert team of diagnosis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients admitted to women health hospital, Assiut university, Assiut
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Model for percise diagnosis of placenta accreta spectrum Using 2d and/or 3d ultrasound doppler to assess: Placental site | (gestational age 28wk-full term) till operation
Model for percise diagnosis of placenta accreta spectrum Using 2d and/or 3d ultrasound doppler to assess: placental thickness | (gestational age 28wk- full term) till operation
Model for percise diagnosis of placenta accreta spectrum Using 2d and/or 3d ultrasound doppler to assess: placental size | (gestational age 28wk- fullterm) till operation
Model for percise diagnosis of placenta accreta spectrum Using 2d and/or 3d ultrasound doppler to assess: placental lacunae | (gestational age 28wk-full term) till operation
Model for percise diagnosis of placenta accreta spectrum Using 2d and/or 3d ultrasound doppler to assess: Loss of placental hypoechoic zone | (gestattional age 28wk-full term) till operation
Model for percise diagnosis of placenta accreta spectrum Using 2d and/or 3d ultrasound doppler to assess: Mean systolic velocity in both uterine arteries | (gestational age 28wks-full term) till time of operation
Model for percise diagnosis of placenta accreta spectrum Using 2d and/or 3d ultrasound doppler to assess: Peak systolic velocity in uteroplacental interface | (gestational age 28wks- full term) till operation
Model for percise diagnosis of placenta accreta spectrum Using 2d and/or 3d ultrasound doppler to assess: Peak systolic velocity in uterovesical interface | (gestational age 28wks- full term) ill operation

SECONDARY OUTCOMES:
precise diagnosis of uterine dehiscence Using 2d and/or 3d ultrasound doppler to assess: Placental site | (gestational age 28wk- fullterm) till operation
precise diagnosis of uterine dehiscence Using 2d and/or 3d ultrasound doppler to assess: Placental size | (gestational age 28wk- full term)till the operation
precise diagnosis of uterine dehiscence Using 2d and/or 3d ultrasound doppler to assess: Placental thickness | (gestational age 28wk-full term) till operation
precise diagnosis of uterine dehiscence Using 2d and/or 3d ultrasound doppler to assess: Placental lacunae | (gestational age 28wk- fullterm) till operation
precise diagnosis of uterine dehiscence Using 2d and/or 3d ultrasound doppler to assess: Loss of placental hypoechoic zone | (gestational age 28wks - fullterm) till operation
precise diagnosis of uterine dehiscence Using 2d and/or 3d ultrasound doppler to assess: Mean systolic velocity in both uterine arteries | (gestational age 28wk- fullterm) till operation
precise diagnosis of uterine dehiscence Using 2d and/or 3d ultrasound doppler to assess: Peak systolic velocity in uteroplacental interface | (gestational age 28wk- fullterm) till operation
precise diagnosis of uterine dehiscence Using 2d and/or 3d ultrasound doppler to assess: Peak systolic velocity in uterovesical interface | (gestational age 28wk-full term) till operation

IPD SHARING:
Plan to Share IPD: No